CLINICAL TRIAL: NCT00544271
Title: Phase IIIb Study to Evaluate Immunogenicity, Antibody Persistency and Reactogenicity of DTPa - INFANRIX and dTpa - BOOSTRIX Vaccines Administered to Healthy Children Previously Primed With 3 Doses of DTPa Vaccine Compared to Placebo (HAVRIX®JUNIOR)
Brief Title: Immunogenicity, Antibody Persistence and Safety of GSK Biologicals' DTPa (INFANRIX) and dTpa (BOOSTRIX) Vaccines.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 263855/035
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Acellular Pertussis; Tetanus; Diphtheria
Keywords: BOOSTRIX; INFANRIX
MeSH Terms: conditions — Tetanus; Diphtheria | interventions — Diphtheria-Tetanus-acellular Pertussis Vaccines; Boostrix; Hepatitis A Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: INFANRIX
Biological: BOOSTRIX
Biological: HAVRIX
  Other Names: INFANRIX; BOOSTRIX

SUMMARY:
To evaluate the immunogenicity, persistence of antibodies and reactogenicity of GSK Biologicals' DTPa (INFANRIX) and dTpa (BOOSTRIX), when administered to subjects 18-20 months old, compared with not giving a booster DTP vaccine at 18-20 months. Study double blinded for the two DTP vaccines and single blinded for the control arm.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children between and including 18 -20 months of age at the time of the vaccination.
* Completed a primary vaccination course with DTPa (INFANRIX) vaccine at 2, 4, and 6 months.
* Written informed consent obtained before study entry from the parents or guardians of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the administration of the study vaccine dose, or planned use during the study period.
* Evidence of previous or intercurrent diphtheria, tetanus, or pertussis disease, or of vaccination against any of these diseases since completion of the primary course of DTPa (INFANRIX) vaccine.

Ages: 18 Months to 20 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 720 (Actual)
Dates: Start 2003-05; Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Anti-diphtheria and anti-tetanus antibody concentration (1M, 15-18M & 27-29M after vacc)
Occurrence of local injection site reactions (1M after vacc).

SECONDARY OUTCOMES:
Antibody concentration to all vaccine antigens (1M, 15-18M & 27-29M after vacc),
Solicited (Day 0-14) & Unsolicited symptoms (Day 0-30),
SAEs (full study).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Carlton, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 263855/035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 263855/035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 263855/035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 263855/035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 263855/035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 263855/035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register